CLINICAL TRIAL: NCT01037439
Title: Comparison of a Modified Adaptive Servoventilation With Conventional Adaptive Servoventilation Processes in Terms of Efficacy Against Complex Nocturnal Breathing Disorders
Brief Title: Comparison of Modified With Conventional Adaptive Servoventilation Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MAEssenASV
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Periodic Breathing; Cheyne-Stokes Respiration
MeSH Terms: conditions — Cheyne-Stokes Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional ASV (Active Comparator): Current adaptive servoventilation therapy algorithm for non invasive ventilation treatment of Cheyne-Stokes Respiration.
  Interventions: Device: Adaptive Servo-controlled Ventilation (ASV)
- Modified ASV (Experimental): Modified adaptive servoventilation algorithm for improved treatment of nocturnal breathing disorders
  Interventions: Device: Adaptive Servo-controlled Ventilation (ASV)

INTERVENTIONS:
Device: Adaptive Servo-controlled Ventilation (ASV) — Pressure support ventilation adapts to meet a target ventilation level that is constantly being assessed
  Other Names: AutoSet CS2; Adapt SV

SUMMARY:
The objective of this study is to compare the modified adaptive servoventilation control algorithm of the with the standardised algorithms of routinely-used servoventilation processes (AutoSet CS2) in terms of the effect on obstructive and central events. The aim is to normalise breathing during sleep and hence eliminate the sleep-related breathing disorder, resulting in even more effective treatment of nocturnal breathing disorders in patients with cardiovascular diseases and sleep apnoea, to ensure optimum therapy success.

DETAILED DESCRIPTION:
Patients with cardiovascular disorders frequently suffer from sleep-related respiratory disorders (SRRD), such as obstructive sleep apnea (OSA) or a specific form of central sleep apnea, Cheyne-Stokes breathing (CSB, periodic breathing). However there is also a significant incidence of complex nocturnal breathing disorders, with both obstructive and central components. Sleep-related breathing disorders of this kind cause decreases in arterial oxygen saturation through brief hypopneas and apneas. Disturbed breathing also causes the patient to wake frequently during the night (arousals), usually during the hyperventilatory phase of CSB. Repeated arousals cause fragmentation of sleep, and therefore a deep sleep deficit. This leads to increased sleepiness during the day and impaired cognitive performance.

Previous studies have shown that Cheyne-Stokes breathing can be treated effectively with adaptive servoventilation. An enhancement to the routinely used algorithm (AutoSet CS2) has been created which allows the algorithm to differentiate between obstructive events and Cheyne-Stokes breathing, and better respond to apneas and hypopneas to eliminate the sleep-related breathing disorder and normalise breathing during sleep.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* consent in writing
* complex nocturnal breathing disorder with Cheyne-Stokes breathing and obstructive sleep apnoea
* AHI > 15/h

Exclusion Criteria:

* acute cardiac decompensation
* acute myocardial infarct within the last 3 months
* post-resuscitation condition within the last 3 months
* post-stroke condition with difficulty in swallowing or persisting hemiparesis
* abuse of medication, alcohol or drugs
* pregnancy
* known to be suffering from a tumour

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Apnea/hypopnea index (AHI) | 1 night sleep
  number of breathing pauses that occur each hour of sleep

SECONDARY OUTCOMES:
Average SaO2 | 1 night sleep
  average percentage of oxygen saturation in the blood
CPAP pressure | 1 night sleep
  Continuous Positive Airway Pressure requirement for elimination of nocturnal breathing disorders
Pressure stability in presence of mask leaks | 1 night sleep
  How much the CPAP pressure varies when mask leak occurs
Minimum SaO2 | 1 night sleep
  The minimum percentage of oxygen saturation recorded in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Teschler, MD, Principal Investigator — University Hospital, Ruhrland Hospital Essen
Locations (1):
- Ruhrland Hospital, Weg, Hesse, Germany